CLINICAL TRIAL: NCT02409914
Title: Brain Metabolism in Women With Polycystic Ovary Syndrome: a PET/MRI Study
Brief Title: Brain Metabolism in Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: 10-153
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2015-04

CONDITIONS: Insulin Resistance
Keywords: Insulin Resistance; Brain metabolism; PET; MRI
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POLYCYSTIC OVARY SYNDROME (PCOS): FDG PET scan,T1-weight MRI and blood were obtained for each participant

SUMMARY:
The purpose of this study is to investigate whether higher insulin resistance in young women with Polycystic ovary syndrome (PCOS) is associated with reduced cerebral metabolic rate of glucose (CMRglu). Brain volumes using magnetic resonance imaging (MRI) and quantitative cerebral glucose uptake using dynamic positron emission tomography (PET) were obtained.

DETAILED DESCRIPTION:
MRI and FDG PET scan for each participant were obtained within an average time frame of 3 weeks. Isulin resistance were assessed with the updated homeostasis model assessment (HOMA2-IR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS
* Age ≤ 35 y
* BMI ≤ 35

Exclusion Criteria:

* Taking medications for diabetes or insulin-sensitizing drugs
* Drug addictions
* Psychiatric illness
* Smoking
* Overt evidence of heart, liver or renal disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with PCOS (n=7) were referred by physician specialist in endocrinology between March, 2010 and September, 2013. The diagnosis of PCOS was based on clinical examination using the Rotterdam criteria.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women with PCOS diagnosed during a clinical examination using the Rotterdam criteria were recruited.
Groups:
- POLYCYSTIC OVARY SYNDROME (PCOS): Women with PCOS. FDG PET scan,T1-weight MRI and a blood sample for the evaluation of insulin resistance were obtained within an average time frame of 3 weeks.
Period: Overall Study
Arm/Group | POLYCYSTIC OVARY SYNDROME (PCOS)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- POLYCYSTIC OVARY SYNDROME (PCOS): Women with PCOS diagnosed during a clinical examination using the Rotterdam criteria.
  PET and MRI exams: FDG PET scan and T1-weight MRI were obtained within an average time frame of 3 weeks.
Arm/Group | POLYCYSTIC OVARY SYNDROME (PCOS)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Global Brain Glucose PET Uptake
Description: Global brain glucose uptake was quantified using FDG with dynamic positron emission tomography.
Time Frame: Single point in time (day 1)
Measure: Mean (Standard Deviation); unit: umol/100 g/min
Groups:
- Polycystic Ovary Syndrome (PCOS): Women with PCOS.
Arm/Group | Polycystic Ovary Syndrome (PCOS)
Number analyzed (Participants) | 7
umol/100 g/min | 34.9 (3.0)

2. Primary Outcome: Brain MR Volumes
Description: T1-weighted brain MR images were obtained on a 1.5 Tesla scanner. Regional volumes were determined using FreeSurfer Suite 5.0 software.
Time Frame: Single point in time (day 2)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Polycystic Ovary Syndrome (PCOS)
Number analyzed (Participants) | 7
ml
  Superior frontal cortex | 22.6 (2.0)
  Supramarginal cortex | 10.3 (1.4)

3. Primary Outcome: Insulin Resistance (HOMA2-IR)
Description: The homeostasis model assessment computational method was used to estimate insulin resistance (HOMA2-IR) from fasting plasma glucose and insulin. The HOMA2-IR is the reciprocal of insulin sensitivity (%S), as a percentage of a normal reference population (normal young adult). A higher score indicates a lower insulin sensitivity.
Time Frame: Single point in time (day 1 during the FDG PET)
Measure: Mean (Standard Deviation); unit: HOMA2-IR score
Arm/Group | Polycystic Ovary Syndrome (PCOS)
Number analyzed (Participants) | 7
HOMA2-IR score | 0.7 (0.3)

ADVERSE EVENTS:
Description: Adverse Events were not monitored/assessed
Arm/Group | POLYCYSTIC OVARY SYNDROME (PCOS)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No